CLINICAL TRIAL: NCT03513744
Title: Evaluation of Nutritional Suitability and Tolerability of a Human Milk Oligosaccharide (HMO) Mix in Infant Formula for Term Infants
Brief Title: Study Evaluating Growth and Tolerance of Infant Formula Containing HMOs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennewein Biotechnologie GmbH (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JEN/008017
Record Dates: First submitted 2018-04-12; First posted 2018-05-02 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Infant Nutrition
Keywords: human milk oligosaccharides; infant formula

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- infant formula containing five HMOs (Experimental)
  Interventions: Dietary Supplement: human milk oligosaccharides
- infant formula (No Intervention)
- breast milk group (No Intervention)

INTERVENTIONS:
Dietary Supplement: human milk oligosaccharides — mixture of five different human milk oligosaccharides
  Arms: infant formula containing five HMOs

SUMMARY:
The primary objective of this clinical study is to investigate the suitability of an infant formula containing five different human milk oligosaccharides to support normal physical growth (evaluated per weight gain), in comparison with infant formula without human milk oligosaccharides, when the formula is fed as the sole source of nutrition.

DETAILED DESCRIPTION:
The main goal of the study is to investigate the suitability of an infant formula containing five different human milk oligosaccharides to support normal physical growth of term infants (evaluated per weight gain, body length and head circumference), in comparison with infant formula without human milk oligosaccharides, when the formula is fed exclusivly in the first four month of life. Additionally, a comparison of the two formula fed groups against a reference group with breastfed infants as well as the WHO growth standard reference tables will be performed. An assessment of safety and tolerability will be performed as well.

As a secondary out come of the study, we will examine the effect of the formula on the infant microbiome, as well as the HMO status of the mother's milk towards the microbial composition of the infant microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* Full-term infant (37 - 42 weeks of gestational age)
* APGAR score of 9 or 10
* Birth weight 2500 - 4500 g

Exclusion Criteria:

* clinically significant condition/ disorder
* Adverse maternal of fetal medical history that may influence growth/development of the subject or tolerance of the infant formula
* readmission to hospital (except for hyperbilirubinemia)
* allergy to cow's milk
* participation in another study

Ages: 1 Day to 13 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
assessment of body weight (in grams) of term infants | 4 month
  growth, assessed by body weight gain, of term infants from enrollment to 4 month of life

SECONDARY OUTCOMES:
assessment of body length (in centimeter) of term infants | 4 month
  growth, assessed as body length, of term infants from enrollment to 4 month of life
assessment of head circumference (in centimeter) of term infants | 4 month
  growth, assessed as head circumference, of term infants from enrollment to 4month of life

OTHER OUTCOMES:
digestive tolerance | 4 month
  stool frequency and consistency
influence of digestion | 4 month
  digestive tolerance parameters ( e.g. rigurgitation, flatulence) will be assessed
influence on behaviour | 4 month
  behavior patterns (e.g.fussiness, cramps, awakings at night) will be assessed
product compliance | 4 month
  intake of infant formula in ml
morbidity | 4 month
  observation of illness
stool microbiota | 4 month
  analysis of the fecal microbiota
HMO composition in breast milk | 4 month
  analysis of HMO composition in mothers breastmilk in the breast-fed arm

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jochum, Dr. med., Principal Investigator — Universitaetsmedizin Berlin, Charité
Locations (9):
- Germany (2):
  - Facharzt für Kinder und Jugendmedizin, Mannheim
  - Klinikum Südstadt Rostock, Rostock
- Italy (2):
  - ASST Spedali Civili di Brescia - Presidio Ospedale dei Bambini, Brescia
  - Ospedale San Raffaele, Milan
- Spain (5):
  - Hospital HM Puerta del Sur, Madrid
  - Hospital HM Monteprincipe, Madrid
  - Hospital HM Nuevo Belen, Madrid
  - Hospital Universitario Sant Joan de Reus, Reus
  - Hospital Joan XXII of Tarragona, Tarragona